CLINICAL TRIAL: NCT03969563
Title: Mindfulness-Based Stress Reduction to Improve Neuropsychological Functioning in Acquired Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D2951-R
Record Dates: First submitted 2019-05-29; First posted 2019-05-31 (Actual); Results first posted 2025-01-22 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Stroke
Keywords: stroke; MBSR; meditation; mindfulness; yoga
MeSH Terms: conditions — Stroke | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: Participants are assigned to either the MBSR or Brain Health education class, in parallel for the duration of the study.
Who Masked: Outcomes Assessor
Masking Description: The neuropsychologist doing the assessments pre- and post-intervention will not be aware of the participant's group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindfulness-based Stress Reduction (MBSR) (Experimental): 8-week Mindfulness-based Stress Reduction class that trains participants in mindfulness, meditation, and yoga.
  Interventions: Behavioral: Mindfulness-based Stress Reduction
- Brain Health Education (Active Comparator): 8-week Brain Health education class that teaches participants about brain-behavior relationships, nutrition, aging facts, sleep, and memory.
  Interventions: Behavioral: Brain Health Education

INTERVENTIONS:
Behavioral: Mindfulness-based Stress Reduction — 8-week Mindfulness-based Stress Reduction class that trains participants in mindfulness, meditation, and yoga.
  Other Names: MBSR
  Arms: Mindfulness-based Stress Reduction (MBSR)
Behavioral: Brain Health Education — 8-week Brain Health education class that teaches participants about brain-behavior relationships, nutrition, aging facts, sleep, and memory.
  Arms: Brain Health Education

SUMMARY:
Thousands of Veterans suffer a stroke every year, and these individuals often suffer emotional and cognitive changes that negatively affect their quality of life as well as their ability to recover. In addition to traditional rehabilitation such as physical and occupational therapy, a number of alternative treatments are now being studied for their ability to enhance patients' recovery following stroke. One of these treatments, Mindfulness-Based Stress Reduction or MBSR, involves an 8-week course that teaches individuals strategies such as breathing techniques, meditation, and movement therapy. The current study proposes to teach MBSR to a group of Veterans with a history of stroke to determine whether this type of intervention has beneficial effects on psychological and cognitive functioning. The investigators hope to find that MBSR is a useful, additional intervention that can improve Veterans' well-being and quality of life as they recover from stroke.

DETAILED DESCRIPTION:
Stroke affects approximately 800,000 Americans every year, including thousands of Veterans, and is a leading cause of disability in the US. While many stroke patients receive rehabilitation during the acute and post-acute phases of stroke, many individuals suffer chronic deficits and have few options for continued treatment. A number of low-cost, alternative treatments are now being tested for their usefulness in treating neuropsychological deficits in chronic stroke patients. One of the best studied of these treatments is Mindfulness-Based Stress Reduction (MBSR), which involves an 8-week course led by a trained instructor. MBSR teaches individuals strategies for coping with their injury, such as meditation, breathing techniques, and yoga. A handful of preliminary studies have shown that MBSR is effective in reducing symptoms of anxiety and depression in stroke patients, as well as enhancing performance on cognitive tasks. However, only a single randomized controlled trial of MBSR in stroke has been published to date, and that study suffered from a number of weaknesses such as the lack of an active control group. Moreover, no previous study has assessed the usefulness of MBSR for stroke in a Veteran population. Therefore, the current study proposes to undertake a rigorous, randomized controlled trial of MBSR in Veterans with a history of stroke, using an active control group, blinded examiners, and a 6-month follow-up session to determine whether the benefits of MBSR are long-lasting. For the study, 120 Veterans with a history of chronic stroke will be recruited: 60 participants will be randomly assigned to the MBSR intervention, and 60 participants will be assigned to a Brain Health class that is matched to the MBSR intervention with respect to the instructor, number of hours of instruction, homework activities, and class size. A blinded examiner will complete a neuropsychological assessment of patients' emotional and cognitive status at three time points: 1) prior to the intervention, 2) following the intervention, and 3) six months later. Evaluation of the MBSR intervention will test for improvements in anxiety and depressive symptomatology following the intervention, relative to the Brain Health group, as well as improvements on a cognitive test battery. It is predicted that improvements associated with the MBSR intervention will still be present at the 6-month follow-up assessment as well. The final objective of the current proposal is to determine whether the site of a patient's stroke plays a role in their ability to benefit from MBSR. Previous research has suggested that left prefrontal cortex plays a critical role underlying the effects of MBSR. Thus, it is predicted that involvement of this brain region will modulate the observed effects. Such information could be used to target those Veterans who can most benefit from the proposed intervention. If shown to be effective, MBSR could provide a low-cost, non-invasive rehabilitative treatment for Veterans with acquired brain injury that can improve their neuropsychological functioning and general sense of well-being. Due to the COVID pandemic, we did not test patients on in-person RBANS cognitive testing as had been originally intended. We also used the Geriatric Depression Scale instead of the Beck Depression Inventory, and the State-Trait Anxiety Inventory instead of the Beck Anxiety Inventory, both of which are highly correlated with each other, due to test availability and cost/copyrights.

ELIGIBILITY:
Inclusion Criteria:

* history of a single, chronic right or left hemisphere stroke

  * defined here as > 3 months post-onset so that residual symptoms have stabilized)
* native English proficiency
* at least mild level of depression

  * 14 on Beck Depression Inventory-II94,95
* and/or mild anxiety

  * 8 on the Beck Anxiety Inventory27
* language within normal limits

  * Western Aphasia Battery score > 93.7104
* scores already available in the investigators' stroke patient database so that language deficits will not interfere with the intervention

Exclusion Criteria:

* a pre-morbid neurologic history or history of schizophrenia spectrum and other psychotic disorders

  * including depressive disorders with psychotic features
* bipolar disorders (to avoid potential confounds in neuropsychological testing)
* Mini-Mental State Examination score <19 (suggesting moderate to severe cognitive impairment that is a contraindication in effectively participating in the MBSR intervention52)
* recent substance abuse/dependence disorder (< 1 year)
* acutely suicidal
* concurrent involvement in another rehabilitation program
* significant visual or hearing disabilities that would preclude participating in the program

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juliana V. Baldo, PhD, Principal Investigator — VA Northern California Health Care System, Mather, CA
Locations (1):
- VA Northern California Health Care System, Mather, CA, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lwi SJ, Paulraj SR, Schendel K, Dempsey DG, Curran BC, Herron TJ, Baldo JV. A Randomized, Controlled Pilot Study of Mindfulness-Based Stress Reduction in Healthy Older Adults. Clin Gerontol. 2023 May-Jun;46(3):330-345. doi: 10.1080/07317115.2022.2137075. Epub 2022 Nov 18. PMID 36398589
- [Derived] Lwi SJ, Chok J, Schendel K, Herron TJ, Curran BC, Baldo JV. A randomized controlled trial of online mindfulness-based stress reduction in chronic stroke. Rehabil Psychol. 2026 Jan 5:10.1037/rep0000651. doi: 10.1037/rep0000651. Online ahead of print. PMID 41490301

RESULTS

PARTICIPANT FLOW:
Groups:
- MBSR: 8-week Mindfulness-based Stress Reduction class that trains participants in mindfulness, meditation, and yoga.
  Mindfulness-based Stress Reduction: 8-week Mindfulness-based Stress Reduction class that trains participants in mindfulness, meditation, and yoga.
Period: Overall Study
Arm/Group | MBSR | Brain Health Education
Started | 57 | 53
Completed | 29 | 30
Not Completed | 28 | 23

BASELINE CHARACTERISTICS:
Population: Of these 57 MBSR and 53 Brain Health Education participants who were enrolled and completed baseline characteristics and were assigned to one of the 2 arms, 36 MBSR and 33 Brain Health participants began the intervention phase of the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | MBSR | Brain Health Education | Total
Number analyzed (Participants) | 57 | 53 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 19 | 36
  >=65 years | 40 | 34 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (7.4) | 67.8 (7.6) | 67.7 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 52 | 52 | 104
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian American | 4 | 0 | 4
  Black | 18 | 10 | 28
  Hispanic/Latine | 4 | 2 | 6
  Native Hawaiian/Pacific Islander | 2 | 2 | 4
  White | 24 | 35 | 59
  Mixed | 5 | 4 | 9
Education [Mean (Standard Deviation); unit: years] | 15 (2.2) | 14.5 (2.8) | 14.8 (2.5)

OUTCOME MEASURES:

1. Primary Outcome: State-Trait Anxiety Inventory
Description: The primary psychological outcome measure is the State-Trait Anxiety Inventory to measure changes in subjective symptoms of anxiety from pre- to post-intervention. The range is 20-80, with 20-37 being no/minimal anxiety and 45-80 being severe anxiety. A lower score post-intervention indicates improvement on this measure.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | MBSR | Brain Health Education
Number analyzed (Participants) | 29 | 30
Score on a scale | 32.8 (9) | 32.5 (11.8)
Statistical Analysis 1: Comparison: MBSR vs Brain Health Education; Test type: Equivalence — Equivalence based on non-significant difference between MBSR and Brain Health groups; p = .694, Mixed Models Analysis; Mean Difference (Final Values) = .3

2. Secondary Outcome: Geriatric Depression Scale - 30
Description: The secondary psychological outcome measure is a change in depression scores from pre- to post-intervention. The range is 0 to 30, with 0 being no/minimal depression and 20-30 being severe depression. A lower score post-intervention indicates improvement on this measure.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | MBSR | Brain Health Education
Number analyzed (Participants) | 29 | 30
Score on a scale | 6.5 (4.5) | 7.9 (6.9)
Statistical Analysis 1: Comparison: MBSR vs Brain Health Education; Test type: Equivalence — Equivalence based on non-significant difference between MBSR vs Brain Health group; p = .837, Mixed Models Analysis; Mean Difference (Final Values) = -1.4

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | MBSR | Brain Health Education
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/53
Other Adverse Events (participants affected / at risk) | 0/57 | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-10-31): https://cdn.clinicaltrials.gov/large-docs/63/NCT03969563/Prot_001.pdf
  • Statistical Analysis Plan (2019-10-31): https://cdn.clinicaltrials.gov/large-docs/63/NCT03969563/SAP_002.pdf
  • Informed Consent Form (2021-08-18): https://cdn.clinicaltrials.gov/large-docs/63/NCT03969563/ICF_000.pdf